CLINICAL TRIAL: NCT04465955
Title: A Phase 2 Multicenter, Randomized, Double-Masked, Sham-Controlled Study of the Safety and Efficacy of Intravitreal Injections of NGM621 in Subjects With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: A Study of NGM621 in Participants With Geographic Atrophy
Acronym: CATALINA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 621-GA-201
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NGM621 Treatment Group A (every 4 weeks) (Experimental): NGM621 single intravitreal (IVT) injection
  Interventions: Biological: NGM621
- NGM621 Treatment Group C (every 8 weeks) (Experimental): NGM621 single IVT injection
  Interventions: Biological: NGM621
- Sham Group B (every 4 weeks) (Sham Comparator): Sham single IVT injection
  Interventions: Other: Sham Comparator
- Sham Group D (every 8 weeks) (Sham Comparator): Sham single IVT injection
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Biological: NGM621 — NGM621 Dose 1
  Arms: NGM621 Treatment Group A (every 4 weeks)
Biological: NGM621 — NGM621 Dose 2
  Arms: NGM621 Treatment Group C (every 8 weeks)
Other: Sham Comparator — Sham Comparator
  Arms: Sham Group B (every 4 weeks); Sham Group D (every 8 weeks)

SUMMARY:
This is a multi-center evaluation of NGM621 in a randomized, double-masked, sham-controlled study in participants with Geographic Atrophy secondary to Age-related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-pregnant, non-lactating) subjects ≥ 55 years
* Standard luminance BCVA score of 34 letters or better using ETDRS charts at the starting distance of 4 meters (approximately 20/200 Snellen equivalent or better) in study eye
* Clinical diagnosis of GA secondary to AMD:

  1. Total GA area must be ≥ 2.5 and ≤ 17.5 mm²
  2. If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm² (0.5 DA), with the overall area of GA ≥ 2.5 and ≤ 17.5 mm²
  3. Well demarcated GA with no anatomical evidence of current or prior CNV in the study eye

Exclusion Criteria:

Study Eye

* GA secondary to a condition other than AMD in either eye (e.g., monogenetic macular dystrophies like Stargardt disease, cone rod dystrophy, or toxic maculopathies)
* Any history of or active choroidal neovascularization (CNV)

Both Eyes

* Any history of or active bacterial, viral, fungal, or parasitic infection in either eye in the 3 months prior to randomization

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals
Locations (65):
- United States (65):
  - Associated Retina Consultants, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Loma Linda University Health, Loma Linda, California
  - University of California Los Angeles, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Institute of California, Palm Desert, California
  - California Eye Specialists, Pasadena, California
  - Retina Consultants San Diego, Poway, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Colorado Retina Associates PC, Golden, Colorado
  - New England Retina Associates PC, Waterford, Connecticut
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - University of Miami, Coral Gables, Florida
  - Specialty Retina Center (Coral Springs), Coral Springs, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Georgia Retina PC, Marietta, Georgia
  - Gailey Eye Clinic - Bloomington, Bloomington, Illinois
  - University of Illinois, Chicago, Illinois
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - Retina Associates, PA, Shawnee Mission, Kansas
  - Thompson Sjaarda, PA, Baltimore, Maryland
  - Elman Retina Group PA, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associated Retina Consultants PC, Royal Oak, Michigan
  - Associated Retina Consultants PC, Traverse City, Michigan
  - Vitreoretinal Surgery PA, Minneapolis, Minnesota
  - Deep Blue Retina Clinical Research, Southaven, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Vitreous Retina Macula Consultants of NY, New York, New York
  - Albany Troy Cataract & Laser Associates, Troy, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Southeast Clinical Research, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - Cascade Medical Research Institute, Springfield, Oregon
  - Eye Care Specialists, Kingston, Pennsylvania
  - Retinovitreous Associates, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Tennessee Retina, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates-Plano, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - University of Virginia, Charlottesville, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Since the study did not meet the study endpoints, there is no plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 320 participants who met all inclusion criteria and no exclusion criteria were randomized to 1 of 4 treatment groups (NGM621 treatment or sham comparator administered either every 4 weeks or every 8 weeks) at 65 sites in the United States. Participants were randomized to 1 of the 4 treatment groups in a ratio of 2 (NGM621 Q4W):1 (Placebo Q4W):2 (NGM621 Q8W):1 (Placebo Q8W).
Groups:
- NGM621 Q4W: Participants who were randomized to a single intravitreal (IVT) injection of 15 mg of NGM621 every 4 weeks (Q4W).
- NGM621 Q8W: Participants who were randomized to a single intravitreal (IVT) injection of 15 mg of NGM621 every 8 weeks (Q8W).
- Sham Q4W+Q8W: Participants who were either randomized to a single intravitreal (IVT) injection of sham comparator every 4 weeks (Q4W) or every 8 weeks (Q8W). As prespecified in the protocol, the sham comparator groups were pooled for analysis purposes.
Period: Overall Study
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Started (Randomized to treatment) | 108 | 105 | 107
Received Treatment | 108 | 104 | 106
Completed | 93 | 89 | 93
Not Completed | 15 | 16 | 14
Not completed — Withdrew consent | 6 | 10 | 7
Not completed — Adverse Event | 6 | 5 | 1
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Other | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Demographic characteristics were assessed in the modified Intent-to-Treat population.
Groups:
- Total: Total of all reporting groups
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W | Total
Number analyzed (Participants) | 108 | 104 | 106 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.5 (8.17) | 79.1 (7.51) | 77.6 (8.42) | 78.4 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 63 | 68 | 198
  Male | 41 | 41 | 38 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 2 | 3
  Black or African American | 0 | 0 | 1 | 1
  Multiple | 1 | 0 | 0 | 1
  Other | 0 | 1 | 1 | 2
  White | 107 | 102 | 101 | 310
Region of Enrollment [Number; unit: participants]
  United States | 108 | 104 | 106 | 318

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Change From Baseline in Geographic Atrophy (GA) Lesion Area
Description: The rate of change from baseline in GA lesion area was measured by a non-invasive imaging technique called fundus autofluorescence (FAF) over the 52 weeks of treatment. FAF refers to the spontaneous emission of light by certain substances within the eye when exposed to a specific wavelength of light and involves quantifying the area and progression of atrophic lesions. The minimal GA lesion area is zero, the maximal GA lesion area is unknown. The higher the GA lesion area, the worse the visual outcome.
Time Frame: Baseline to Week 52
Population: The rate of change from baseline in the GA lesion area was assessed in the modified Intent-to-Treat population.
Measure: Mean (Standard Error); unit: mm^2 per year
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 108 | 104 | 106
mm^2 per year | 2.243 (0.138) | 2.237 (0.140) | 2.393 (0.138)
Statistical Analysis 1: Comparison: NGM621 Q4W vs Sham Q4W+Q8W; Rate of Change Difference Between NGM621 Q4W and Pooled Sham; Test type: Superiority; p = 0.4345, Random coefficient model; Covariates included terms for time, treatment-by-time interaction, baseline fellow eye CNV status, baseline focality, and baseline GA lesion location; Mean Difference (Final Values) = -0.150, 95% CI 2-sided [-0.528 to 0.227]
Statistical Analysis 2: Comparison: NGM621 Q8W vs Sham Q4W+Q8W; Rate of Change Difference Between NGM621 Q8W and Pooled Sham; Test type: Superiority; p = 0.4217, Random coefficient model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.155, 95% CI 2-sided [-0.536 to 0.225]

2. Primary Outcome: Number of Participants With Ocular Treatment-emergent Adverse Events in the Study Eye
Description: A treatment-emergent adverse event (TEAE) was an adverse event (AE) that occurred during or after the first dose of study treatment.
Time Frame: Baseline to end of study (Week 56)
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 108 | 104 | 106
Participants
  Any TEAE | 57 | 51 | 49
  Any Treatment-related TEAE | 6 | 5 | 1
  Any Serious TEAE | 8 | 8 | 3
  Any TEAE Leading to Treatment Discontinuation | 0 | 1 | 0
  Any Sight Threatening TEAE | 6 | 6 | 3
  Any Severe TEAE | 1 | 3 | 0

3. Secondary Outcome: The Change From Baseline in Geographic Atrophy (GA) Lesion Area
Description: Geographic atrophy lesion area was measured by a non-invasive imaging technique called fundus autofluorescence (FAF). FAF refers to the spontaneous emission of light by certain substances within the eye when exposed to a specific wavelength of light and involves quantifying the area and progression of atrophic lesions. The minimal GA lesion area is zero, the maximal GA lesion area is unknown. The higher the GA lesion area, the worse the visual outcome.
Time Frame: Baseline up to Week 52
Population: The change from baseline in GA lesion area was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 90 | 89 | 90
mm^2 | 2.172 (1.5026) | 2.235 (1.4203) | 2.479 (1.4028)

4. Secondary Outcome: The Rate of Change From Baseline in the Square Root of Geographic Atropy (GA) Lesion Area
Description: Geographic atrophy lesion area was measured by fundus autofluorescence (FAF). FAF refers to the spontaneous emission of light by certain substances within the eye when exposed to a specific wavelength of light and involves quantifying the area and progression of atrophic lesions.
Time Frame: Baseline up to Week 52
Population: The rate of change from baseline in the square root of GA lesion area was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: mm^2 per year
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 90 | 89 | 90
mm^2 per year | 0.389 (0.2352) | 0.388 (0.2200) | 0.423 (0.2225)

5. Secondary Outcome: The Change From Baseline in Best Corrected Visual Acuity Score
Description: Best Corrected Visual Acuity Score is the best possible vision an eye can achieve with corrective lenses, typically glasses or contact lenses. BCVA was assessed by the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. ETDRS letter score is calculated when >20 letters are read correctly at 4.0 meters; the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters plus 30. If <20 letters are read correctly at 4.0 meters, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters (number of letters recorded on line 1.0), plus the total number of letters in the first six lines read correctly at 1.0 meter. Therefore, the ETDRS letter score could result in a score of 0-100, where lower scores indicate better vision.
  The change from baseline in BCVA is being report with negative scores indicating an improvement in vision.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Best Corrected Visual Acuity Score was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 88 | 85 | 88
score on a scale | -2.7 (9.55) | -5.6 (12.80) | -2.7 (9.71)

6. Secondary Outcome: The Change From Baseline in Low Luminance Visual Acuity Score
Description: Low Luminance Visual Acuity Score measures vision in low-light conditions. It was assessed by the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters.
  ETDRS letter score is calculated when >20 letters are read correctly at 4.0 meters; the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters plus 30. If <20 letters are read correctly at 4.0 meters, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters (number of letters recorded on line 1.0), plus the total number of letters in the first six lines read correctly at 1.0 meter. Therefore, the ETDRS letter score could result in a score of 0-100, where lower scores indicate better vision.
  A lower (negative) LLVA score compared to baseline indicates a decline in visual acuity. A higher (positive) LLVA score compared to baseline indicates an improvement in visual acuity.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Low Luminance Visual Acuity Score was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 92 | 88 | 88
score on a scale | 0.1 (12.38) | -1.4 (12.45) | -2.31 (13.00)

7. Secondary Outcome: The Change From Baseline in Low Luminance Deficit Score
Description: Low Luminance Deficit (LLD) Score was assessed by the Early Treatment of Diabetic Retinopathy Study (ETDRS) letters at a starting distance of 4 meters. ETDRS letter score is calculated when >20 letters are read correctly at 4.0 meters; the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters plus 30. If <20 letters are read correctly at 4.0 meters, the visual acuity letter score is equal to the total number of letters read correctly at 4.0 meters (number of letters recorded on line 1.0), plus the total number of letters in the first six lines read correctly at 1.0 meter. Therefore, the ETDRS letter score could result in a score of 0-100, where lower scores indicate better vision.
  A LLD is the difference between standard visual acuity and LLVA, with a LLD >13 ETDRS letters suggesting potential visual abnormality. The change from baseline in LLD is being report with negative scores indicating an improvement in vision.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Low Luminance Deficit Score was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 92 | 88 | 88
score on a scale | -2.9 (13.48) | -5.3 (16.16) | -0.5 (14.10)

8. Secondary Outcome: The Change From Baseline in Average Binocular Reading Speed
Description: Average binocular reading speed was assessed by Minnesota Low-Vision Reading Test (MNRead) or Radner reading charts. The change from baseline in average binocular reading speed is reported with a higher (positive) reading speed (wpm) indicates better reading ability, while a lower (negative) reading speed indicates poorer reading ability.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Binocular Reading Speed was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: words per minute
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 66 | 58 | 68
words per minute | -9.17 (39.154) | -16.90 (36.853) | -8.70 (39.844)

9. Secondary Outcome: The Change From Baseline in Binocular Critical Print Size
Description: Binocular critical print size was assessed by the Minnesota Low-Vision Reading Test (MNRead) or Radner reading charts. MNRead uses a logarithmic scale (LogMAR) to represent print sizes, with each step representing a 0.1 LogMAR difference. The chart ranges from +1.3 LogMAR (equivalent to 20/400 at 40 cm) to -0.5 LogMAR (equivalent to 20/6 at 40 cm). The change from baseline in binocular critical print size is being reported with a higher (positive) LogMAR value for critical print size indicating that a person needs larger print sizes to maintain their maximum reading speed, while a lower (negative) LogMAR value indicates that they can read smaller print sizes at their maximum speed.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Binocular Critical Print Size was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 66 | 58 | 68
logMAR | -0.01 (0.290) | -0.01 (0.334) | 0 (0.280)

10. Secondary Outcome: The Change From Baseline in Binocular Reading Acuity
Description: Binocular reading acuity was assessed by the Minnesota Low-Vision Reading Test (MNRead) or Radner reading charts. MNRead uses a logarithmic scale (LogMAR) to represent print sizes, with each step representing a 0.1 LogMAR difference. The chart ranges from +1.3 LogMAR (equivalent to 20/400 at 40 cm) to -0.5 LogMAR (equivalent to 20/6 at 40 cm). Binocular reading acuity is the smallest print size (in LogMAR) that a person can read easily and accurately. The change from baseline in binocular reading acuity is being reported with a higher LogMAR value for reading acuity indicates poorer reading ability, while a lower LogMAR value indicates better reading ability.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Binocular Reading Acuity was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 79 | 79 | 80
logMAR | 0.047 (0.2760) | 0.086 (0.2812) | 0.058 (0.2455)

11. Secondary Outcome: The Change From Baseline in Functional Reading Independence Index Composite Score
Description: The Functional Reading Independence (FRI) Index Composite Score is a 7-item patient questionnaire developed to evaluate the effect of geography atrophy on a patient's ability to independently perform reading activities. The FRI Index yields mean scores ranging from 1-4, with 1=unable to do and 4=totally independent. The FRI Index composite score is calculated by averaging the item-level scores across the seven questions, higher sores indicate better FRI. The change from baseline in FRI is being reported with lower (negative) values indicating a decline in FRI.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Functional Reading Independence Index was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 91 | 88 | 90
score on a scale | -0.14 (0.597) | -0.15 (0.512) | -0.20 (0.675)

12. Secondary Outcome: The Change From Baseline in National Eye Institute Visual Functioning Questionnaire Composite Score
Description: The National Eye Institute Visual Functioning Questionnaire Composite Score is calculated by averaging the scores of the 11 vision-targeted subscales, excluding the general health rating question, on a scale of 0 to 100, with higher scores indicating better vision-related function. The change from baseline is being reported with a negative value indicating a decline in vision function.
Time Frame: Baseline up to Week 52
Population: The change from baseline in National Eye Institute Visual Functioning Questionnaire was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 91 | 88 | 91
score on a scale | -1.97 (11.075) | -3.74 (10.024) | -2.96 (11.549)

13. Secondary Outcome: The Change From Baseline in Systemic Complement Activity (CH50)
Description: Systemic Complement Activity is a blood test that measures the overall activity of the complement system, a group of proteins crucial for the immune system's function. Low CH50 levels can be associated with certain infections. CH50 levels of 41 to 90 hemolytic units per mL (U/mL) is considered normal. The change from baseline in CH50 is being reported.
Time Frame: Baseline up to Week 52
Population: The change from baseline in Systemic Complement Activity was assessed in participants with available data in the modified Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: units/mL
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 77 | 70 | 75
units/mL | 18.16 (51.339) | 24.17 (56.244) | 26.595 (54.077)

14. Secondary Outcome: Number of Anti-Drug Antibody (ADA)-Negative Participants
Description: The incidence of anti-drug antibody (ADA) was assessed in serum.
Time Frame: Baseline up to Week 52
Population: ADA-negative participants were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
Number analyzed (Participants) | 93 | 86 | 85
Participants | 93 | 86 | 85

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening, baseline, Week 1 and every 4 weeks thereafter up to end of study (Week 56).
Description: As prespecified in the protocol, the sham comparator groups were pooled for analysis purposes.
Arm/Group | NGM621 Q4W | NGM621 Q8W | Sham Q4W+Q8W
All-Cause Mortality (participants affected / at risk) | 4/108 | 2/104 | 2/106
Serious Adverse Events (participants affected / at risk) | 32/108 | 24/104 | 29/106
Other Adverse Events (participants affected / at risk) | 33/108 | 34/104 | 31/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NGM621 Q4W (N=108) | NGM621 Q8W (N=104) | Sham Q4W+Q8W (N=106)
Dry age-related macular degeneration (Eye disorders) | 4 | 4 | 3 — Includes fellow eye serious TEAEs: N=1 NGM621 Q8W and N=2 Sham (Q4W+Q8W)
Visual acuity reduced (Eye disorders) | 2 | 3 | 0
Visual impairment (Eye disorders) | 1 | 2 | 1
Retinal artery occlusion (Eye disorders) | 1 | 1 | 0
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0 | 0 — Only reported in fellow eye
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 — Only reported in fellow eye
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 3
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NGM621 Q4W (N=108) | NGM621 Q8W (N=104) | Sham Q4W+Q8W (N=106)
Conjunctival haemorrhage (Eye disorders) | 14 | 14 | 8
Visual acuity reduced (Eye disorders) | 5 | 8 | 6
Dry age-related macular degeneration (Eye disorders) | 7 | 5 | 7
Visual impairment (Eye disorders) | 5 | 7 | 4
Retinal haemorrhage (fellow eye) (Eye disorders) | 2 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT04465955/Prot_SAP_000.pdf